CLINICAL TRIAL: NCT02307136
Title: Evaluation of the Impact of Within-hospital Trajectories of Patients Admitted in Intensive Care Units (ICU) From Emergency Departments
Acronym: SUREA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI11013-AOR11114
Record Dates: First submitted 2014-11-27; First posted 2014-12-04 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Intensive Care Units; Emergency Department
Keywords: intensive care units; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter cohort aims to assess the impact of within-hospital trajectories of patients admitted in intensive care units from emergency departments on vital prognosis of patients, duration of hospital stay and hospital costs.

As secondary objectives, the study will:

* assess the impact of clinical and demographic characteristics on hospital trajectories of patients.
* assess the impact of emergency units workload, beds availability in medical units and in intensive care units, and global hospital organisation on patients care trajectories.

DETAILED DESCRIPTION:
The study will be performed in emergency departments and ICUs of university hospitals. 15 emergency departments and 36 ICUs of APHP (the public hospital system of the city of Paris) will be involved.

The study will assemble the data from 50,000 to 80,000 patients in total.

Eligible patients are admitted in ICUs between 01/01/2007 and 12/31/2011.

Extraction of the patients' data will be performed with processing software utilised in APHP, i.e. Healthcare Information System Program (PMSI, Urqual, Gilda...etc.).

Collected patients' data span the period from admission in emergency department or medical department unitl hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient directly admitted in ICU from emergency departments of APHP (the public hospital system of the city of Paris).
* Adult patient indirectly transferred to ICU from an hospitalization unit, initially admitted from an emergency department of APHP.

Exclusion Criteria:

* Patient transferred from APHP toward an external hospital, outside APHP, before being admitted in an ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population under study is formed of patients admitted in 3 types of intensive care units (Medical intensive care unit, Surgical Intensive Care Unit and Cardiac Intensive Care Unit), transferred from emergency departments, either directly, or from another Department such as a Unit of short durations of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mortality | throughout the study: 5 years
  Mortality in ICU and in other hospital units
Rate of direct transfer | throughout the study: 5 years
  Rate of direct transfer from Emergency Unit to ICU
Rate of indirect transfer | throughout the study: 5 years
  Rate of indirect transfer from a hospitalization Unit to ICU
Duration of stay in emergency department, in ICU and in hospital | throughout the study: 5 years
  Duration of stay in emergency department, in ICU and in hospital
Mode of discharge from ICU | throughout the study: 5 years
  Mode of discharge from ICU and direction of patient (home, other structures etc.)

SECONDARY OUTCOMES:
Severity scores | throughout the study: 5 years
  Severity scores in ICU
Use and duration of mechanical ventilation | throughout the study: 5 years
  Use and duration of mechanical ventilation for patient during ICU stay
Score of burden of care in ICU | throughout the study: 5 years
  Score of burden of care in ICU
Percentage of patients with ICU stay | throughout the study: 5 years
  Percentage of patients with ICU stay
Percentage of patients with continuing care | throughout the study: 5 years
  Percentage of patients with continuing care after discharge from the ICU
Frequency of dialysis | throughout the study: 5 years
  Frequency of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Enrique CASALINO, MD, PhD, Principal Investigator — APHP
Locations (1):
- Emergency Department, Bichat-Claude Bernard Hospital, Paris, Île-de-France Region, France